CLINICAL TRIAL: NCT01241201
Title: A Study Proposal to Investigate the Sequels of Mucosal Inflammation Caused by ETEC Infection - the Effects of Probiotics.
Brief Title: Intestinal Barrier Function and Probiotics.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: VSL Pharmaceuticals (Industry); NIZO Food Research (Other)
Responsible Party: Ministry of Health, Welfare and Sport
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: P9067
Record Dates: First submitted 2010-10-29; First posted 2010-11-16 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Intestinal Permeability; Challenge Test; Intestinal Health; Inflammation
Keywords: intestinal health; probiotics; inflammation; biomarkers
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo (Placebo Comparator): placebo for probiotic treatment
  Interventions: Dietary Supplement: Priobiotic supplement VSL#3

INTERVENTIONS:
Dietary Supplement: Priobiotic supplement VSL#3 — four weeks, twice daily two sachets of VSL#3, a priobitics mixture

SUMMARY:
Rationale: Enterotoxigenic Escherichia coli (ETEC) bacteria adhere to the mucosa of the proximal intestines. There it produces an toxin which presents a local and relevant challenge to the intestines. This is proposed to give an indication of general resistance and/or the local resistance of the intestines. The sequel of events of mucosal inflammation will be characterized in this study. In addition we will evaluate the effects of probiotics by comparing the infection symptoms and by measuring faecal weight and mucus in faeces.

Objective: The main objective of this study is to investigate the effect of probiotics on the sequels of ETEC administration as intestinal permeability, inflammation and clinical signs as total faecal output, relative faecal dry weight and mucin excretion in faeces. In addition, the sequels of the mucosal inflammation will be characterized and biomarkers will be searched.

DETAILED DESCRIPTION:
Study population: 36 Healthy male volunteers; age >= 21 and <= 40 years. Intervention: One group receives twice daily two sachets containing 450 billion live freeze-dried lactic acid bacteria per sachet and the other group receives twice daily two placebo sachets.

Study design: The study is designed as a randomized, parallel, placebo-controlled, double-blind study. Study substance (probiotics) and placebo will be given during 4 weeks.

Main study parameters/endpoints: The main study parameter is the percent change in faecal dry weight and total faecal output between the probiotics group and the placebo group. In addition, intestinal permeability, inflammation and other clinical symptoms will be evaluated.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In this study healthy male volunteers will be challenged with an attenuated ETEC strain after three weeks of either probiotics or placebo. This infection will lead to a mild traveller's diarrhoea in the subjects during approximately three days maximally. Sequels of this infection and the effects of commercially available probiotics compared to placebo will be followed up. The subjects will therefore collect their faeces on several days, record their defecation pattern and gastro-intestinal complaints during four weeks, undergo a physical examination and five venapunctions, and visit our facilities in total on 8 days (excluding two pre-study visits). The oral administration of probiotics in a healthy population is not associated with risk.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the

   * health and lifestyle questionnaire, (P9067 F02; in Dutch)
   * physical examination
   * results of the pre-study laboratory tests
2. Males, Age >= 21 and <= 40 years at Day 01 of the study
3. Body Mass Index (BMI) >= 20 and < 33 kg/m2. Preferably in high and low body fat mass ranges as to be determined by waist circumference
4. Normal Dutch eating habits as assessed by P9067 F02
5. Voluntary participation
6. Having given written informed consent
7. Willing to comply with the study procedures, including the ETEC challenge
8. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years
9. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned.

Exclusion Criteria:

Subjects with one or more of the following characteristics will be excluded from participation:

1. Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalatory administration of substances
3. Having a history of medical or surgical events that may significantly affect the study outcome, including gastrointestinal illness or surgical operations,
4. Use of antibiotics, immunosuppressive drugs, antacids, laxatives or anti-diarrhoeal drugs in the last 3 months before the study
5. Alcohol consumption > 28 units/week for males
6. Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening
7. Reported slimming or medically prescribed diet
8. Reported vegan, vegetarian or macrobiotic
9. Not willing to be off working as a food handler, in child care or as a healthcare worker with direct patient contact during the week of ETEC contamination
10. Not willing to give up blood donation during the study.
11. Personnel of TNO Quality of Life, their partner and their first and second degree relatives
12. Not having a general practitioner
13. Not willing to accept information-transfer concerning participation in the study, or information regarding his/her health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Faecal weight and mucus (diarrhoea) | day 01
  Characteristics of the faeces will be determined (% wet and dry weight)
Faecal weight and mucus (diarrhoea) | day 20
  Characteristics of the faeces will be determined (% wet and dry weight)
Faecal weight and mucus (diarrhoea) | day 22
  Characteristics of the faeces will be determined (% wet and dry weight)
Faecal weight and mucus (diarrhoea) | day 23
  Characteristics of the faeces will be determined (% wet and dry weight)
Faecal weight and mucus (diarrhoea) | day 24
  Characteristics of the faeces will be determined (% wet and dry weight)

SECONDARY OUTCOMES:
intestinal permeability | day 01, 20 and day 22
  Determine the intestinal permeability before and after probiotic supplementation and especially after infection of the intestines.

CONTACTS AND LOCATIONS:
Overall Officials: W J Pasman, PhD, Principal Investigator — TNO
Locations (1):
- TNO Quality of Life, Zeist, Utrecht, Netherlands

REFERENCES:
- [Background] Bovee-Oudenhoven IM, Lettink-Wissink ML, Van Doesburg W, Witteman BJ, Van Der Meer R. Diarrhea caused by enterotoxigenic Escherichia coli infection of humans is inhibited by dietary calcium. Gastroenterology. 2003 Aug;125(2):469-76. doi: 10.1016/s0016-5085(03)00884-9. PMID 12891550